CLINICAL TRIAL: NCT05847348
Title: A Prospective, Open-Label, Single-Arm, Multi-center Study to Evaluate the Diagnostic Efficacy and Safety of 68Ga-PSMA-11 PET/CT or PET/MRI in Patients With Biochemical Recurrent Prostate Cancer
Brief Title: 68Ga-PSMA-11 Efficacy in Detecting BCR Prostate Cancer in Chinese Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Grand Pharmaceutical (China) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-PSMA-11-001
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Biochemical Recurrence of Malignant Neoplasm of Prostate; Prostate Cancer; BCR Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: This study aims to recruit 110 prostate cancer patients with elevated PSA (BCR) after radical prostatectomy or radical radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (68Ga-PSMA-11) (Experimental): 111 ~ 259 MBq 68Ga-PSMA-11 will be administered intravenously to participants over 3- 5 minutes.
  After 50-100 minutes post 68Ga-PSMA-11 injection, participants will be scanned (PET/CT or PET/MRI) from the mid-thigh to the apex of the skull. Participants will be placed in a supine position with the arms raised overhead.
  Interventions: Drug: 68Ga-PSMA-11; Other: PET/CT or PET/MRI

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — A single dose of 111 - 259 MBq administered intravenously over 3 -5 minutes
  Other Names: Illucix; gallium Ga 68 Gozetotide
Other: PET/CT or PET/MRI — PET/CT or PET/MRI will be acquired no sooner than 50 minutes post injection and not later than 100 minutes post injection with 68Ga-PSMA-11
  Other Names: Imaging by PET

SUMMARY:
This is a prospective, open-label, single-arm, multicenter bridging study in Chinese patients with prostate cancer. This multicenter study is planned to be conducted in patients with biochemical recurrence (BCR) of elevated PSA after radical prostatectomy or radical radiotherapy. This study investigates how well 68Ga-PSMA-11 PET/CT works in detecting BCR prostate cancer in Chinese patient. 68Ga-PSMA-11, developed by Telix, is a new molecular entity tracer with the trade name Illuccix®, which is approved by FDA for the examination of: 1) patients with suspected metastatic PC who are scheduled for initial treatment; 2) patients with biochemical recurrence of elevated PSA levels after initial radical radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to understand and provide written informed consent document.
2. Are Chinese males aged ≥ 18 years.
3. Have histopathologically confirmed prostate adenocarcinoma and have undergone radical prostatectomy and/or radical radiotherapy and experienced biochemical recurrence (PSA should be measured within 30 days of screening).

   1. Post radical prostatectomy (RP) PSA ≥0.2 ng/mL measured 6 weeks after RP
   2. Post radiation therapy - ASTRO-Phoenix consensus definition Nadir + ≥ 2 ng/mL rise in PSA;
4. Have a Karnofsky performance status ≥ 60 (or ECOG/WHO equivalent).
5. Agree to practice a highly effective method of contraception for at least 28 days after 68Ga-PSMA-11 administration.
6. Are willing and able to comply with scheduled

Exclusion Criteria:

1. Have a prior history of any other malignancy within the last year, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.
2. Have prior use of radionuclides with an interval of less than 10 physical half-lives before the administration of 68Ga-PSMA-11.
3. Are participating or plan to participate in any drug or device clinical study during the study period.
4. Have a known hypersensitivity to the active ingredient or its components of 68Ga-PSMA-11.
5. Cannot lie flat or remain still while a PET scan is being performed or cannot tolerate a PET scan.
6. Have prior history of salivary gland disease or Paget's disease.
7. Have a history of fracture and anemia within the last year.
8. Have abnormalities in physical examination, ECG, and protocol-specified clinical laboratory tests during the Screening Period that, in the judgment of the investigator, could affect safety or compliance.
9. Is deemed not suitable for participating in this trial in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is limited to males only
Enrollment: 110 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of 68Ga-PSMA-11 PET/CT or PET/MRI for detection of tumour on a patient level confirmed by histopathology/biopsy, clinical (PSA) and conventional imaging follow-up. | 12 months
  The PPV [PPV (%) = TP* /(TP + FP**)] will be determined by the combination of histopathology/biopsy and conventional imaging and/or PSA follow-up results as the true criteria (composite criteria) and the results observed by 68Ga-PSMA-11 PET (positive/negative).

SECONDARY OUTCOMES:
Incidence of adverse events | 3 days
  Safety will be reported descriptively as rates of patient reported adverse events. Additionally, adverse events will be characterized and quantified by Common Terminology Criteria for Adverse Events
Clinical management in biochemical recurrence patients. | 3 days
  The impact of 68Ga-PSMA-11 PET/CT or PET/MRI on clinical management in biochemical recurrence patients will be assessed through the completion of Medical Management Questionnaires completed prior to and after 68Ga-PSMA-11 PET/CT or PET/MRI.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - West China Hospital of Sichuan University, Sichuan
  - Wuhan Union Hospital, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Affiliated Hosptial of Jiangnan University, Wuxi

IPD SHARING:
Plan to Share IPD: No